CLINICAL TRIAL: NCT02973672
Title: A Phase I Study Assessing the Safety and Performance of SGM-101, a Fluorochrome-labeled Anti-carcino-embryonic Antigen Monoclonal Antibody for the Detection of Neoplastic Lesions in Patients With Colorectal Cancer or Pancreatic Cancer
Brief Title: Phase I of SGM-101 in Patients With Cancer of the Colon, Rectum or Pancreas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Surgimab (Industry)
Collaborators: Centre for Human Drug Research, Netherlands (Other); Leiden University Medical Center (Other); Erasmus Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SGM-CLIN02
Record Dates: First submitted 2016-11-16; First posted 2016-11-25 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Colon Cancer; Rectum Cancer; Pancreas Cancer; Metastatic Colorectal Cancer; Recurrent Colorectal Carcinoma
Keywords: Fluorescence; Surgery; Cancer; SGM-101; Near Infrared; Immunophotodetection
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGM-101 (Experimental)
  Interventions: Drug: SGM-101

INTERVENTIONS:
Drug: SGM-101 — 4 days before surgery, SGM-101 will be administered to the patient by intravenous injections.
  Other Names: SGM 101; SGM101

SUMMARY:
This study evaluates the safety and performance of SGM-101, a Carcinoembryonic Antigen (CEA)-specific chimeric antibody conjugated with a NIR emitting fluorochrome, for the visualization of CEA-expressing cancers during surgery. SGM-101 is injected 2 to 4 days before surgery and visualized using an optimized camera system.

DETAILED DESCRIPTION:
Surgery is the most important therapy for patients with cancer of the colon, rectum or pancreas. Complete resection, which is a crucial factor in the prognosis of a patient, is challenging as surgeons have to rely on visual appearance and palpation to discriminate between tumor and normal tissue.

Carcinoembryonic antigen (CEA) is a tumor-specific marker that is highly expressed in a number of tumors of epithelial origin (such as colorectal carcinoma and pancreas carcinoma) while it is minimally expressed in normal adult tissues. The compound that will be studied in this research project is SGM-101, a CEA-specific chimeric antibody conjugated with a near-infrared (NIR) emitting moiety. The hypothesis is that, following preoperative iv administration of SGM-101 in patients with carcinoma of the colon, rectum or pancreas, SGM-101 will bind to CEA expressing cancer cells and these cells can then be visualized with a NIR fluorescence imaging system, thereby increasing the chance of radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old;
* Patient should be scheduled and eligible for surgery because of a clinical diagnosis of cancer of the colon, rectum or cancer of the pancreas;
* Both pancreatic and colorectal cancer patients: Circulating plasma CEA ≥ the upper limit of normal range (eg ≥ 3.0 ng / ml);
* Patient suffering from recurrences and metastasis of colorectal cancer: Rising circulating plasma CEA
* Patients should be capable and willing to give informed consent before study specific procedures.

Exclusion Criteria:

* Anticancer therapy (e.g. chemotherapy, radiotherapy (except for routine pre-operative radiotherapy for colorectal cancer), targeted therapy, concomitant systemic immune therapy, or any experimental therapy) within 4 weeks before inclusion;
* History of a clinically significant allergy;
* Circulating plasma concentration CEA ≥ 300 ng / ml;
* Other malignancies either currently active or diagnosed in the last 5 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma;
* Patients pregnant or breastfeeding (pregnancy should be ruled out by an assay of βhCG plasma within 4±1 weeks prior to administration of the conjugate), lack of effective contraception in male or female patients with reproductive potential;
* Laboratory abnormalities defined as:

Colorectal cancer patients only:

* Aspartate AminoTransferase, Alanine AminoTransferase, Gamma Glutamyl Transferase) or Alkaline Phosphatase levels above 5 times the or;
* Total bilirubin above 2 times the Upper Limit Normal (ULN) or; Both pancreatic and colorectal cancer patients:
* Serum creatinine above 1.5 times the ULN or;
* Absolute neutrophils counts below 1.5 x 109/L or;
* Platelet count below 100 x 109/L or;
* Hemoglobin below 4 mmol/L (females) or below 5 mmol/l (males);
* Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections;
* Any condition that the investigator considers to be potentially jeopardizing the patients' wellbeing or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-01; Primary Completion 2019-04-15 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events | up to 10 days after the surgery
  An Adverse Event (AE) is any untoward medical occurrence in a subject who is participating in a clinical study performed. The adverse event does not necessarily have to follow the administration of a study drug, or to have a causal relationship with the study drug. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory or vital sign finding), symptom, or disease temporally associated with the study participation, whether or not it is related to the study drug.

SECONDARY OUTCOMES:
Tumor-to-background ratio (TBR) for fluorescence | day 4
Serum SGM-101 concentrations | up to 1 month after surgery
  Individual serum SGM-101 concentrations will be plotted versus time per individual using both a linear and log y-axis. Additionally, concentration versus time curves will be plotted per treatment group as a spaghetti plot.
  Concentrations will be summarized by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander L Vahrmeijer, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (3):
- Netherlands (3):
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center Cancer Institute, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lwin TM, Hoffman RM, Bouvet M. The future of tumour-specific fluorescence-guided surgery for pancreatic cancer. Lancet Gastroenterol Hepatol. 2020 Aug;5(8):715-717. doi: 10.1016/S2468-1253(20)30123-0. Epub 2020 May 14. No abstract available. PMID 32416765
- [Derived] Schaap DP, de Valk KS, Deken MM, Meijer RPJ, Burggraaf J, Vahrmeijer AL, Kusters M; SGM-101 study group. Carcinoembryonic antigen-specific, fluorescent image-guided cytoreductive surgery with hyperthermic intraperitoneal chemotherapy for metastatic colorectal cancer. Br J Surg. 2020 Mar;107(4):334-337. doi: 10.1002/bjs.11523. Epub 2020 Jan 21. PMID 31960953
- [Derived] Boogerd LSF, Hoogstins CES, Schaap DP, Kusters M, Handgraaf HJM, van der Valk MJM, Hilling DE, Holman FA, Peeters KCMJ, Mieog JSD, van de Velde CJH, Farina-Sarasqueta A, van Lijnschoten I, Framery B, Pelegrin A, Gutowski M, Nienhuijs SW, de Hingh IHJT, Nieuwenhuijzen GAP, Rutten HJT, Cailler F, Burggraaf J, Vahrmeijer AL. Safety and effectiveness of SGM-101, a fluorescent antibody targeting carcinoembryonic antigen, for intraoperative detection of colorectal cancer: a dose-escalation pilot study. Lancet Gastroenterol Hepatol. 2018 Mar;3(3):181-191. doi: 10.1016/S2468-1253(17)30395-3. Epub 2018 Jan 30. PMID 29361435